CLINICAL TRIAL: NCT01426997
Title: Phenotyping Major Depression With Increased Inflammation
Brief Title: Phenotype Depression Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Psychiatry and Behavioral Sciences, Emory University
Other Study IDs: IRB00039107; 1R01MH087604-01A1 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Diurnal plasma samples are collected hourly from 9 am to 9 pm once; Cerebrospinal fluid once; mRNA from peripheral blood leuckocytes collected 5 times; DNA for analysis of genetic polymorphisms is collected once.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- High inflammation group (CRP>3 mg/L): Forty-five participants each with a diagnosis of major depressive disorder and a CRP level >3 mg/L
- Medium inflammation group (CRP=1-3 mg/L): Forty-five participants each with a diagnosis of major depressive disorder and a CRP level = 1-3 mg/L
- Low inflammation group (CRP<1 mg/L).: Forty-five participants each with a diagnosis of major depressive disorder and a CRP level <1 mg/L

SUMMARY:
To facilitate the development of a personalized approach to the treatment of patients with major depression, this study is designed to elaborate the clinical and neurobiological phenotype of depressed patients with increased inflammation. The data obtained in this proposal will allow the investigators to test the hypothesis that depression and inflammation interact to elaborate a relatively discreet phenotype that warrants an individualized approach to diagnosis and treatment of patients with depression. Moreover, the identification of specific environmental risk factors for inflammation will foster the elaboration of preventative strategies for patients at risk.

DETAILED DESCRIPTION:
One hundred and thiry-five patients with major depression diagnosed based on DSM-IV TR criteria between the ages of 21 and 65 (males, females and minorities) will be recruited. Forty-five patients with high inflammation as defined by a CRP >3 mg/L will be enrolled along with 45 depressed patients with medium inflammation (CRP=1-3mg/L) and 45 depressed patients with low inflammation (CRP<1mg/L) will complete a 2 night inpatient stay in Emory University Hospital's research unit, the Atlanta Clinical and Translational Science Institute (ACTSI). Participants will undergo psychiatric and neurocognitive assessments, sleep studies and blood and cerebral spinal fluid (CSF) sampling.

ELIGIBILITY:
Inclusion Criteria:

* age 21-65 years including males, females and minorities
* diagnosis of DSM-IV major depression or Bipolar I or II with current episode of depression
* HDRS-17 > 20 and HDRS-24 > 24
* negative pregnancy test for women of childbearing potential
* not breast feeding
* stable on current dose of psychotropic medication or free from all psychotropic medications for 4 weeks prior to EUH CIN admission (8 weeks for fluoxetine)
* no suicide attempt within six months of screening

Exclusion Criteria:

* evidence of untreated or poorly controlled endocrine, cardiovascular, pulmonary, hematological, renal, or neurological disease
* history of CNS trauma or active seizure disorder requiring medication unless otherwise approved by principle investigator
* autoimmune or inflammatory disorder of any kind
* chronic infection (e.g. hepatitis B or C or HIV)
* chronic use of agents known to affect the immune system including glucocorticoid therapy within the past 1 year, methotrexate within the past 1 year, chemotherapy of any kind (past or present), immunotherapy of any kind (past or present), aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) (within the past 2 weeks) and statins (within the past 1 month) unless otherwise approved by principle investigator
* hemoglobinopathies (e.g. thalassemia)
* a positive pregnancy test
* organ transplants
* cancer of any type
* a score of <28 on the Mini Mental Status Exam (MMSE)unless otherwise approved by principle investigator
* meets criteria for schizophrenia (Given overlap of generalized anxiety disorder (GAD) with major depression, GAD will not be exclusionary)
* current eating disorders
* active abuse of alcohol or illicit/prescription drugs within the past year unless otherwise approved by principle investigator.
* MGH-S >3 unless otherwise approved by principle investigator
* BMI >40 unless otherwise approved by the principle investigator
* active suicidal intent or plan and a score >2 on the HDRS suicide item (item #3).
* any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and thiry-five patients with major depression diagnosed based on DSM-IV TR criteria between the ages of 21 and 65 (males, females and minorities) will be recruited. Forty-five patients with high inflammation as defined by a CRP >3 mg/L will be enrolled along with 45 depressed patients with medium inflammation (CRP=1-3mg/L) and 45 depressed patients with low inflammation (CRP<1mg/L)
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2010-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
We are using clinician administered and self report psychiatric measurements to compare relevant symptom domains in patients with major depression and increased inflammation versus patients with major depression without increased inflammation. | Inpatient visit
  Behavior: Hamilton Depression Rating Scale (HAM-D); Inventory of Depressive Symptoms-Self Report (IDS-SR); Salpetriere Retardation Rating Scale (SRRS); Snaith-Hamilton Pleasure Scale (SHAPS); Multidimensional Fatigue Inventory (MFI); Neuropsychology: Finger tapping task; Reaction Time Task (CANTAB); Trial Making Test, Part A; Digit Symbol Test; Stocking of Cambridge

SECONDARY OUTCOMES:
We are measuring immune markers for the identification of relevant immunologic patterns of activation in patients with major depression and increased inflammation versus patients with major depression without increased inflammation. | Inpatient visit; Day #2
  Immune Markers: plasma and CSF IFN-alpha, IL-6, sIL-6R, TNF-alpha, sTNFR 1 and 2, IL-1 beta, IL-1ra, sIL-2R and MCP-1; PBMC mRNA expression of genes with responsive elements for NF-kB and MAPK gene expression as well as intracellular phosphorylated p38 as determined by flow cytometry; polymorphisms in genes encoding for IL-1, IL-6, TNF-alpha (and their soluble receptors) as well as MCP-1

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Psychiatry and Behavioral Sciences, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No